CLINICAL TRIAL: NCT04929678
Title: A Prospective, Multi-Center Study of the Braive™ Growth Modulation System When Used in the Treatment of Pediatric Patients Diagnosed With Juvenile or Adolescent Idiopathic Scoliosis
Brief Title: Study of the Braive Growth Modulation System for Progressive Pediatric Scoliosis
Acronym: BRAIVE IDE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Spinal and Biologics (Industry)
Collaborators: Medical Metrics Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT19009SD1901; 287046 (Other: IRAS)
Record Dates: First submitted 2021-05-24; First posted 2021-06-18 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Juvenile Idiopathic Scoliosis; Adolescent Idiopathic Scoliosis
Keywords: Juvenile Idiopathic Scoliosis; Adolescent Idiopathic Scoliosis; Progressive Scoliosis; BRAIVE; Anterior Vertebral Body Tethering; AVBT; Growth modulation system

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Braive™ Growth Modulation System (Braive™ GMS) (Experimental)
  Interventions: Device: Braive™ Growth Modulation System (Braive™ GMS)

INTERVENTIONS:
Device: Braive™ Growth Modulation System (Braive™ GMS) — The Braive™ GMS is designed as a growth-modulation, non-fusion technique, which utilizes patients' remaining growth potential to limit further progression of the curve, to provide correction of the thoracic spine, and allow continued growth while maintaining mobility.
  The system consists of the following components: Braid, Fixed Angle Screws (FAS), Plate, and Break-Off Set Screw.

SUMMARY:
The purpose of this study was to establish probable benefits and evaluate the safety and preliminary effectiveness of the Braive™ GMS when used in the treatment of pediatric progressive scoliosis.

ELIGIBILITY:
Inclusion Criteria:

A subject must meet all of the following inclusion criteria to participate in this study:

* Has a diagnosis of juvenile or adolescent idiopathic scoliosis
* Is skeletally immature with a Sanders Score of ≥2 to ≤5
* Has failed conservative care as per investigator's assessment
* Has a main thoracic Cobb angle between 30 and 60 degrees
* Has a Lenke Classification of 1A, 1B, or 1C
* Has kyphosis ≤ 40 degrees with a sagittal thoracic modifier N or negative
* Informed Consent Form/Assent and Authorization to Use and Disclose Health Information (if applicable) have been signed by Parent/legal guardian and/or patient/participant per local requirement.

Exclusion Criteria:

A subject will be excluded from participating in this study for any of the following reasons:

* Has undergone previous spinal fusion procedure(s) at the affected levels
* Is pregnant or plans to become pregnant within the first 24-months of the study
* Has a curve that requires instrumentation below L1
* Has spinal MRI abnormalities (e.g., CHIARI malformation, Syrinx greater than 4mm, tethered cord)
* Has any type of non-idiopathic scoliosis
* Has a left-sided curve
* Has an associated syndrome
* Has a history of malignant hyperthermia
* Has an active or significant risk of infection (immunocompromised)
* Has inadequate tissue coverage over the operative site as per investigator's assessment
* Has a suspected or documented allergy or intolerance to implant materials
* Has a major psychiatric disorder / history of drug abuse that would interfere with the subject's ability to comply with study instructions or might confound the study interpretation as per investigator's assessment (DSM-5 can be used as a reference)
* Is a ward of the court/state
* Has had prior ipsilateral or contralateral chest surgery
* Has severe chronic lung disease (e.g., asthma, bronchiectasis)
* Has poor bone quality, as determined by the investigator, that may limit anterior fixation
* Is unwilling or unable to return for follow-up visits and/or follow intra-operative and/or postoperative instructions
* Concurrent participation in another clinical study that may add additional safety risks and/or confound study results

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-08-12 (Actual); Primary Completion 2025-04-11 (Actual); Study Completion 2029-12-25 (Estimated)

PRIMARY OUTCOMES:
Summary of device-related adverse events up to 24 months | Baseline to 24 months.
  Device related adverse events are any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, related to the investigational medical device whether anticipated or unanticipated.
  Summary will be based on both Investigators and Medtronic relatedness assessment.

SECONDARY OUTCOMES:
Assessment of procedure-related adverse events up to 24 months | Baseline to 24 months.
  Procedure related adverse events are any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, related to the procedure.
  Summary will be based on both Investigators and Medtronic relatedness assessment.
Assessment of secondary Spinal surgeries related to the original study device up to 24 months. | Baseline to 24 months and up to skeletal maturity
  Some adverse events or treatment failures may lead to additional surgical interventions. Relatedness of these subsequent spinal surgical interventions will be assessed Total events and total number of subjects who have additional surgeries will be summarized. The numbers of revisions (total, preventive and non-preventive), removals, reoperations and other surgeries will also be summarized.
  A relatedness determination will be made by the investigator to the original study device and the original study surgery to a subsequent surgical intervention.
Assessment of device deficiency up to 24 months | Baseline to 24 months and up to skeletal maturity
  A device deficiency (DD) is an inadequacy of a medical device with respect to its identity, quality, durability, reliability, safety or performance. Device deficiencies include malfunctions, use errors, and inadequate labeling.
Change from baseline in main thoracic Cobb angle at all available postoperative time points | Baseline, immediately after the surgery, 3, 6, 12, 18, 24 months, and annually until skeletal maturity is reached.
  Main Thoracic Cobb Angle will be calculated from the PA (posteroanterior) TL (thoracic/lumbar) spine radiograph. Main Thoracic Cobb Angle is reported in units of degrees. A positive angle indicates a curve where the apex is to the subject's right of the adjacent vertebra, i.e. the angle opens to the subject's left. A negative angle indicates a curve where the apex is to the subject's left of the adjacent vertebra, i.e., the angle opens to the subject's right.
Change from baseline in proximal thoracic Cobb angle at all available postoperative timepoints | Baseline, immediately after the surgery, 3, 6, 12, 18, 24 months, and annually until skeletal maturity is reached.
  Proximal Thoracic Cobb Angle will be calculated from the PA TL spine radiograph. The Proximal Thoracic Cobb Angle is reported in units of degrees.
Change from baseline in thoracolumbar/lumbar Cobb angle at all available postoperative timepoints | Baseline, immediately after the surgery, 3, 6, 12, 18, 24 months, and annually until skeletal maturity is reached.
  Thoracolumbar/Lumbar Cobb Angle will be calculated from the PA TL spine radiograph. Thoracolumbar/Lumbar Cobb Angle will be reported in units of degrees.
Change from post-op baseline in Instrumented Cobb Angle at all available postoperative time points. | Immediately after the surgery, 3, 6, 12, 18, 24 months, and annually until skeletal maturity is reached.
  The Instrumented Cobb Angle will be calculated from the PA TL Spine radiograph. It will be measured by drawing lines through the superior endplate of the upper instrumented vertebra and the inferior endplate of lower instrumented vertebra. The Instrumented Cobb Angle upper and lower end vertebrae will be defined at PostOp and maintained for all follow-up measurements. Instrumented Cobb Angle will be reported in units of degrees.
Change from baseline in thoracic kyphosis at all available postoperative timepoints | Baseline, immediately after the surgery, 3, 6, 12, 18, 24 months, and annually until skeletal maturity is reached.
  Thoracic Kyphosis will be calculated from the Lateral TL Spine radiograph and will be measured as the angle between the superior endplate of T5 and the inferior endplate of T12. Thoracic Kyphosis is reported in units of degrees. Positive angle corresponds to kyphotic curvature, whereas negative angle corresponds to lordotic curvature.
Change from baseline in Lumbar Lordosis at all available postoperative timepoints. | Baseline, immediately after the surgery, 3, 6, 12, 18, 24 months, and annually until skeletal maturity is reached.
  Lumbar Lordosis will be calculated from the Lateral TL Spine radiograph and will be measured as the angle between the superior endplate of S1 and the superior endplate of T12. Lumbar Lordosis is reported in units of degrees. Negative angle corresponds to lordotic curvature, and positive angle corresponds to kyphotic curvature.
Change from baseline in coronal balance at all available postoperative timepoints. | Baseline, immediately after the surgery, 3, 6, 12, 18, 24 months, and annually until skeletal maturity is reached.
  Coronal Balance will be measured from the PA TL Spine radiograph. . A vertical line is drawn down from the center of the C7 vertebral body (C7PL), and a vertical line is drawn up from the center of the superior endplate of S1 (also known as the center sacral vertical line; "CSVL"). The distance between these lines is recorded in units of millimeters. The sign is positive if C7PL falls to right of the CSVL and negative if it falls to the left as viewed on the PA image.
Change from baseline in Sagittal Balance at all available postoperative timepoints | Baseline, immediately after the surgery, 3, 6, 12, 18, 24 months, and annually until skeletal maturity is reached.
  Sagittal Balance will be measured from the Lateral TL Spine radiograph. A vertical line is drawn down from the center of the C7 vertebral body (also known as the Sagittal C7 plumb line, "Sagittal C7PL"), and a vertical line drawn from the posterior-superior corner of S1. The distance between these lines is recorded in units of millimeters. The sign is positive if the plumb line falls anterior to the posterior-superior corner of S1 and negative if it falls posterior.
Change from baseline in total vertical thoracic spine height (T1-T12) at all available postoperative timepoints. | Baseline, immediately after the surgery, 3, 6, 12, 18, 24 months, and annually until skeletal maturity is reached.
  Total Vertical Thoracic Spine Height will be calculated from the PA TL Spine radiograph. Total Vertical Thoracic Spine Height is defined as the vertical distance between the level of the midpoint of the superior endplate of T1 and the midpoint of the inferior endplate of T12 and will be reported in units of centimeters.
Change from baseline in total vertical spine height (T1-S1) at all available postoperative timepoints | Baseline, immediately after the surgery, 3, 6, 12, 18, 24 months, and annually until skeletal maturity is reached.
  Total Vertical Spine Height will be calculated from the PA TL Spine radiograph. Total Vertical Spine Length is defined as the vertical distance between the level of the midpoint of the superior endplate of the T1 superior endplate and the midpoint of the superior endplate of S1 and will be reported in units of centimeters.
Change from baseline in Scoliosis Research Society-22 Patient Questionnaire (SRS-22) at all available postoperative timepoint | Baseline to 3, 6, 12, 18, 24 months, and annually until skeletal maturity is reached.
  The SRS-22 contains 22 questions covering 5 domains: function/activity 5 items; pain 5 items; self-perceived image 5 items; mental health 5 items; and satisfaction with treatment 2 items. Each item is scored from 1 (worst) to 5 (best). Each domain has a total sum score ranging from 5 to 25, except for satisfaction, which ranges from 2 to 10. The sum of the first 4 domains gives a maximum subtotal of 100, and when the satisfaction domain is included, the maximum total is 110. Higher score means better outcome.
Status of return to full activity within 3 months per Scoliosis Research Society-22 Patient Questionnaire (SRS-22) | 3 months.
  SRS-22's subdomain function/activity will be utilized to evaluate the status of return to full activity. The subdomain has 5 items and will be scored on a scale from 1 (worst) to 5 (best). Higher score means better outcome.

CONTACTS AND LOCATIONS:
Locations (4):
- Mayo Clinic, Rochester, Minnesota, United States
- Canada (2):
  - IWK Health Centre, Halifax, Nova Scotia
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
- The Newcastle upon Tyne Hospitals NHS Foundation Trust - Royal Victoria Infirmary, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: No